CLINICAL TRIAL: NCT03625869
Title: First Randomized Study of Pressure-controlled Intermittent Coronary Sinus Occlusion (PiCSO) in Acute Myocardial Infarction
Brief Title: Pressure-controlled Intermittent Coronary Sinus Occlusion (PiCSO) in Acute Myocardial Infarction
Acronym: PiCSO-AMI-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Miracor Medical SA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIR-CIP 0002
Record Dates: First submitted 2018-08-03; First posted 2018-08-10 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: STEMI; Anterior MI
Keywords: PiCSO; PiCSO Impulse System
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Anterior Wall Myocardial Infarction

STUDY DESIGN:
Intervention Model Description: A prospective, multicenter, randomized (1:1), controlled, study
Who Masked: Outcomes Assessor
Masking Description: Analysis of the primary endpoint, infarct size 5-days post MI assessed by CMR, will be analyzed by an independent Corelab, blinded to the allocated treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): This is the actual control group receiving conventional therapy, ie. percutaneous coronary intervention.
- PICSO (Experimental): This arm will be treated with Pressure controlled intermittent Coronary Sinus Occlusion (PiCSO) in addition to conventional therapy (percutaneous coronary intervention).
  Interventions: Device: PiCSO

INTERVENTIONS:
Device: PiCSO — After blood flow restoration, the subjects meeting all inclusion and none exclusion criterial will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes (at minimum 30 minutes) whereas the treatment should be continued during and post stent insertion, but should not exceed a maximum duration of 90 minutes. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed.
  Arms: PICSO

SUMMARY:
The objective of this study is to assess efficacy and safety of Pressure-controlled intermittent Coronary Sinus Occlusion (PiCSO) therapy started post flow restoration but prior to stenting during percutaneous coronary intervention (PCI) compared to standard PCI in the setting of acute ST-segment elevation anterior myocardial infarction (STEMI).

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized (1:1), controlled, study. Patients with an ST-segment elevated anterior infarct eligible for PCI will be invited to participate in the PiCSO-AMI-I study. After consent as per pproved ethics committee requirements, baseline assessments will be performed. PCI of the culprit vessel should be performed per standard practices. After blood flow restoration, the subjects meeting all inclusion and none exclusion criterial will be enrolled into the study and randomized either to PiCSO Group or Control Group. If the subject is randomized to PiCSO Group, the coronary sinus (CS) will be cannulated through the femoral vein and the PiCSO Impulse Catheter will be placed in the CS. In the event the PiCSO Impulse Catheter cannot be placed in the CS within 30 minutes, the physician should proceed with the regular PCI and the PiCSO treatment will be considered a failure. Once PiCSO Impulse Catheter is placed into CS, PiCSO treatment is started followed by stenting. The physician shall target a PiCSO treatment of 45 minutes (at minimum 30 minutes) whereas the treatment should be continued during and post stent insertion, but should not exceed a maximum duration of 90 minutes. At the end of the PiCSO treatment, the PiCSO Impulse Console is stopped and the PiCSO Impulse Catheter is removed. The patient is seen for a FU visit at 5 days, 30 days, 6 months, 1 year, 2 year and 3 years post index procedure. 5 days and 6 months post index the patient will get a CMR scan. At every FU visit safety data and health status will be documented and quality of life questionnaire will be completed.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Culprit lesion in proximal or mid LAD
3. Pre-PCI TIMI flow 0 or 1.
4. Symptoms onset time consistent with myocardial ischemia (e.g. persistent chest pain, shortness of breath, nausea/vomiting, fatigue, palpitations or syncope) ≤ 12 h.
5. ECG evidence of acute anterior myocardial infarction with ST-elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous anterior precordial ECG leads (one of which should be V2, V3, or V4) in men or ≥ 1.5 mm (0.15 mV) in women
6. Patient is deemed eligible for primary PCI
7. STEMI patients: consent as per approved national ethical committee specific requirements prior to the procedure.

Exclusion criteria:

1. Implants or foreign bodies in the coronary sinus
2. Known allergy to polyurethanes, PET or stainless steel
3. Known pregnancy and breastfeeding
4. Pericardial effusion (cardiac tamponade)
5. Central hemodynamically relevant left/right shunt
6. Previous MI or CABG
7. History of stroke, TIA or reversible ischemic neurological deficit within last 6 months
8. Known coagulopathy
9. Need for circulatory support or pre-procedural ventilation
10. Patients with cardio-pulmonary resuscitated (CPR) cardiac arrest for more than 5 minutes
11. Patient not suitable for femoral vein access
12. Contraindication to cardiac magnetic resonance imaging (CMR), e.g. claustrophobia, foreign body implants incompatible with CMR, gadolinium intolerance.
13. Active participation in another drug or device investigational study
14. Known severe kidney disease or on hemodialysis
15. Unconscious on presentation
16. Patients under judicial protection, legal guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Infarct size 5 days post MI | 5 days post MI
  Difference in myocardial infarct size (extent of myocardial necrosis quantified by delayed gadolinium enhancement presented as a percentage of LV mass) between the PiCSO Group and the Control Group, assessed by CMR at 5 days post index PCI

SECONDARY OUTCOMES:
Infarct size 6 months post MI | 6 months post MI
  Myocardial infarct size (% of LV mass) assessed by CMR at 6 months post index PCI
MVO | 5 days post MI
  Occurrence and extent of microvascular obstruction (MVO, % of LV mass) and hemorrhage assessed by CMR at 5 days post index PCI
LVEF | 5 days and 6 months post MI
  LVEF assessed by CMR at 5 days and 6 months post index PCI
LVESV | 5 days and 6 months post MI
  LVESV assessed by CMR at 5 days and 6 months post index PCI
LVEDV | 5 days and 6 months post MI
  LVEDV assessed by CMR at 5 days and 6 months post index PCI
Myocardial Salvage | 5 days and 6 months post MI
  Myocardial Salvage Index at 5 days and 6 month post index PCI
ST-segment resolution | 90 minutes
  ST-segment resolution at 90 minutes post flow restoration
Device and Procedural success, assessed as percent of subjects with successful access, delivery, and retrieval of the device and its delivery system | 1 day
  Device success and procedural success rate presented as % of subjects

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Banning, Prof., Principal Investigator — Study principal Investigator
Locations (17):
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Odense University Hospital, Odense
- France (3):
  - CHU Hôpiteaux de Bordeaux, Hôpital Haut Lévéque, Bordeaux
  - Centre Hospitalier Régional Universitaire de Lille, Lille
  - Centre Hospitalier Universitaire de Toulouse, Toulouse
- Klinikum Coburg GmbH, Coburg, Germany
- Pauls Stradins Clinical University Hospital, Riga, Latvia
- Switzerland (2):
  - Bern University Hospital, Bern
  - EOC Ospedale Regionale di Lugano - Civico, Lugano
- United Kingdom (8):
  - Golden Jubilee National Hospital, Clydebank
  - New Edinburgh Royal Infirmary, Edinburgh
  - Royal Brompton and Harefield Hospital, Harefield
  - Leeds Teaching Hopsitals, Leeds
  - Liverpool Heart and Chest Hospital, Liverpool
  - St Bartholomew's Hospital, London
  - Freeman Hospital, Newcastle
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Maria GL, Greenwood JP, Zaman AG, Carrie D, Coste P, Valgimigli M, Behan M, Berry C, Erglis A, Panoulas VF, Van Belle E, Juhl Terkelsen C, Hunziker Munsch L, Jain AK, Lassen JF, Palmer N, Stone GW, Banning AP. Pressure-Controlled Intermittent Coronary Sinus Occlusion (PiCSO) in Acute Myocardial Infarction: The PiCSO-AMI-I Trial. Circ Cardiovasc Interv. 2024 Apr;17(4):e013675. doi: 10.1161/CIRCINTERVENTIONS.123.013675. Epub 2024 Apr 16. PMID 38626079